CLINICAL TRIAL: NCT02179385
Title: Coaching for Health to Achieve New Goals in Empowerment for Diabetes
Brief Title: Empowerment and Support for the Diabetic Patient
Acronym: CHANGE-D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clalit Health Services (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Margalit (Margita) Goldfracht, Department Manager of Quality Promotion, Community Medical Division, Clalit Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0130-13-COM
Record Dates: First submitted 2014-06-25; First posted 2014-07-01 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Type II diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- Health coaching (Experimental): Patients receive health coaching via the phone, face to face or group support, according to patients' choice
  Interventions: Behavioral: Health Coaching
- Standard of Care (Placebo Comparator)

INTERVENTIONS:
Behavioral: Health Coaching
  Arms: Health coaching

SUMMARY:
CHANGE-D objectives are to evaluate to what extent personal coaching for healthy lifestyle and treatment adherence improves clinical outcomes among uncontrolled diabetic patients.

Evaluate to what extent personal coaching for healthy lifestyle and treatment adherence improves self treatment among uncontrolled diabetic patients.

DETAILED DESCRIPTION:
Research Group 300 type 2 diabetics: 150 from Jewish sector and 150 from Arab sector will be recruited from 7-10 clinics in each district: North District and Haifa District A personal coaching intervention will be tailored from the offered tools: Face to face, group, telephone Participants will be monitored for clinical and self treatments outcomes Comparison Group 300 patients with similar characteristics to the research group will receive Clalit's standard of care Participants will be monitored for clinical and self treatments outcomes like the research group

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* At least one oral anti diabetic drug
* HbA1c above 7.5% ot above 0.5% of personal target
* Preparedness for change
* Fluent Hebrew or Arabic

Exclusion Criteria:

* Type 1 diabetes
* Pregnancy or lactation
* Incompetency to sign consent
* Participation in another clinical trial
* Unstable psychotic disease
* Complex health condition

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Clinical composite | 0, 6, 12, 18 months from randomization
  Change from baseline in a composite endpoint of HbA1c, BMI, Blood Pressure, Lipids at 6, 12 and 18 months from randomization

SECONDARY OUTCOMES:
Change in Self Treatment Score | 0, 6, 12, 18 months from randomization
  Change from baseline in Self treatment diabetes questionnaire score at 6, 12 and 18 months from randomization
Change in Self Efficacy Score | 0, 6, 12, 18 months from randomization
  Change from baseline in Self Efficacy questionnaire score at 6, 12 and 18 months from randomization

OTHER OUTCOMES:
Change in Quality of life score | 0, 12 months from randomization
  Change from baseline in Diabetes Quality of Life questionnaire score at 12 months from randomization